CLINICAL TRIAL: NCT00263536
Title: Pilot Program for Targeted Prevention of Child or Adolescent Weight Gain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 060039; 06-CH-0039
Record Dates: First submitted 2005-12-08; First posted 2005-12-08 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2016-08-16

CONDITIONS: Overweight Adolescents; Overweight
Keywords: Obesity; Adiposity; Binge Eating; Social Functioning; Eating Disorders; Prevention; Adolescence; Adolescent Weight Gain; Overweight
MeSH Terms: conditions — Overweight; Obesity; Bulimia; Social Adjustment; Feeding and Eating Disorders | interventions — Interpersonal Psychotherapy

INTERVENTIONS:
Procedure: Interpersonal Psychotherapy

SUMMARY:
This study will examine whether family-based interpersonal psychotherapy (FB-IPT) is an effective tool for helping pre-adolescent girls and boys at risk for become obese to reduce weight gain. IPT is a time-limited group therapy for preventing and treating depression in children. It is also effective for treating binge eating disorder in adults and has resulted in weight maintenance or modest weight loss in obese adults. IPT focuses on improving how people relate to one another by relating symptoms to personal problem areas and then developing strategies for dealing with these problems. Girls and boys between the ages of 8-13 years of age who are in good general health with the exception of being overweight and whose body mass index (BMI) is above the 85th percentile for their age and sex may be eligible for this study. Candidates are screened with a physical examination, measurement of their height and weight, blood and urine tests, a DEXA scan (x-ray scan that measures body fat, muscle and bone mineral content), and questionnaires and an interview to obtain information about the child's general health, social and psychological function, and eating patterns. Parents are also screened for their health and are asked to give blood samples for genetic studies and participate in a few questionnaires and interviews.

Participants are randomly assigned to participate in FB-IPT or a health education program. Both programs involve 12 weekly visits. At the end of the study, the body weight and mood of the girls and boys in both groups are compared.

Participants (a parent and their child) meet individually with the therapist for 12 sessions (each approximately an 45 minutes ). Girls and boys offered FB-IPT have meetings in which they develop strategies for dealing with the problems girls struggle with that may lead to increased eating. Girls and boys in the health education group have meetings that focus on teaching teens children to live healthier lives and review topics related to developing and maintaining healthy eating and exercise.

All participants are evaluated at the end of the 12-week program and asked to return to the NIH for follow-up visits at post treatment, 6 and 12 months following initiation of the program.

Each child and parent will be compensated for their time and inconvenience with $40 for completing all pre-program assessments, $40 for attending the 12 week follow-up visit, $40 for the 6 month follow-up visit, and $40 for the 1-year follow-up. Therefore, each child may receive up to $160, and the participating parent may receive up to $160. If a child's second biological parent is also willing to give a genetic sample and undergo interviews, the second parent can also receive $40 for a single visit to the NIH.

DETAILED DESCRIPTION:
The most prevalent disordered eating pattern described in overweight youth is loss of control (LOC) eating, during which individuals experience an inability to control the amount of food they are consuming. LOC eating is associated cross-sectionally with greater adiposity in children and adolescents, and appears to predispose youth to gain weight or body fat above that expected due to normal growth, thus likely contributing to obesity in susceptible individuals. No prior studies have examined whether LOC eating can be decreased by interventions in children or adolescents, or whether programs reducing LOC eating affect weight gain. Interpersonal Psychotherapy (IPT), a form of psychotherapy that has been adapted for the treatment of eating disorders, has demonstrated efficacy in reducing binge eating episodes and inducing modest weight losses (or at least weight stabilization) among adults diagnosed with binge eating disorder. In Study 1, we proposed a pilot study of the efficacy of group IPT as an intervention to slow the trajectory of weight gain in 36 overweight or at-risk for overweight youth who report symptoms of LOC eating. We hypothesized that reductions in LOC eating among adolescents who engage in such episodes and who are at risk for obesity will decrease the likelihood of inappropriate weight gain. In this pilot study, changes in body composition of adolescent girls participating in a 12-week IPT group intervention were compared with those of girls participating in a health education program at 6 month and 1 year follow-up visits. Significantly more girls who participated in IPT stabilized their weight compared to girls who participated in health education. These promising preliminary data were the basis for an adequately powered trial of adolescent IPT for the prevention of excessive weight gain that is currently underway (NICHD Protocol 08-CH-0139). In Study 2, we wish to pilot an excess weight gain prevention program targeting LOC eating behaviors in middle childhood youth and in their parents. In Study 2 the prevention programs will be delivered in a parent-child dyadic format instead of an adolescent group format. Enrolling children and their parents will also allow pilot exome sequencing genetic analyses to be conducted.

ELIGIBILITY:
* INCLUSION CRITERIA:

Volunteers will qualify if they meet the following criteria:

* Good general health. A normal history and physical examination with the exception of overweight will be required.
* Age greater than or equal to 12 and < 18 years at the start of the study.
* Female.
* Body mass index measured at the NIH is within the 75th 97th percentile for age, gender, and race.
* English speaking.
* Ability to complete study procedures including the ability to participate in a group.

Individuals will be individually assessed to determine their suitability for group treatment. School placement (e.g. special education) will be used as an estimate of cognitive functioning.

- As assessed by the Eating Disorder Examination structured clinical interview (see methods), a history of LOC eating (objective or subjective bulimic episodes, or both) or no reports of LOC eating.

EXCLUSION CRITERIA:

Volunteers will be excluded (and referred to non-experimental treatment programs as needed) for the following reasons:

* Presence of major illnesses: renal, hepatic, gastrointestinal, most endocrinologic (e.g., Cushing syndrome, hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication). Nonserious medical illnesses, such as seasonal allergies, will be reviewed on a case-bycase basis.
* Presence of an obesity-related medical complication that would require a more aggressive weight loss intervention approach. Such comorbidities include hyperlipidemia (LDL-cholesterol > 130 mg/dL), hypertension (defined by age- sexand height- specific standards (115) fasting hyperglycemia (fasting glucose > 126 mg/dL) and nonalcoholic steatohepatitis (ALT above NIH Clinical Center laboratory norms with consistent radiologic findings and absence of another cause such as infectious hepatitis).
* Regular use of prescription medications. Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting study medication. Individuals taking medications for most conditions will be excluded, but medication use for non-serious conditions (e.g., acne) will be considered on a caseby- case basis. In particular, participants currently prescribed SSRI s, neuroleptics, tricyclics, stimulants, or any medication known to affect body weight or eating will be excluded.
* Current involvement in psychotherapy or a structured weight loss program,
* Weight loss during the past 2 months for any reason exceeding 3% of body weight.
* Pregnant or recently pregnant girls (within 1 year of delivery).
* History of an eating disorder or a current eating disorder (other than binge eating disorder) as determined by medical history or if uncovered during the study s structured clinical interviews. Subjects found to have an eating disorder other than binge eating disorder at baseline will be referred to mental health specialists for further evaluation and treatment.
* Current pregnancy or breast feeding. A negative pregnancy test before starting the study will be required. Because pregnancy is a state in which weight gain is expected and appropriate, pregnant individuals would not be suitable for this study. Sexually active females must be using an effective form of birth control. These methods include total abstinence (no sex), oral contraceptives ( the pill ), an intrauterine device (IUD), levonogestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended.
* Individuals who have DSM-IV-TR major depressive disorder, psychoses, current substance or alcohol abuse, conduct disorder, or a diagnosed psychiatric disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study. Individuals whose parents or guardians have current substance abuse or a diagnosed psychiatric disorder or other condition that, in the opinion of the investigators, would impede adherence with the study

Each participant will receive a written explanation of the purposes, procedures, and potential hazards of the study. Communication of this information and of the participant s assent, as well as the consent of the parent or guardian, will be documented in the medical record. All participants will be informed of their right to withdraw from the study.

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 147 (Actual)
Dates: Start 2005-12-05; Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jack A Yanovski, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Hedley AA, Ogden CL, Johnson CL, Carroll MD, Curtin LR, Flegal KM. Prevalence of overweight and obesity among US children, adolescents, and adults, 1999-2002. JAMA. 2004 Jun 16;291(23):2847-50. doi: 10.1001/jama.291.23.2847. PMID 15199035
- [Background] Freedman DS, Khan LK, Dietz WH, Srinivasan SR, Berenson GS. Relationship of childhood obesity to coronary heart disease risk factors in adulthood: the Bogalusa Heart Study. Pediatrics. 2001 Sep;108(3):712-8. doi: 10.1542/peds.108.3.712. PMID 11533341
- [Background] Freedman DS, Khan LK, Serdula MK, Dietz WH, Srinivasan SR, Berenson GS. Inter-relationships among childhood BMI, childhood height, and adult obesity: the Bogalusa Heart Study. Int J Obes Relat Metab Disord. 2004 Jan;28(1):10-6. doi: 10.1038/sj.ijo.0802544. PMID 14652621
- [Derived] Manoli I, Sysol JR, Head PE, Epping MW, Gavrilova O, Crocker MK, Sloan JL, Koutsoukos SA, Wang C, Ktena YP, Mendelson S, Pass AR, Zerfas PM, Hoffmann V, Vernon HJ, Fletcher LA, Reynolds JC, Tsokos MG, Stratakis CA, Voss SD, Chen KY, Brown RJ, Hamosh A, Berry GT, Chen XS, Yanovski JA, Venditti CP. Lipodystrophy in methylmalonic acidemia associated with elevated FGF21 and abnormal methylmalonylation. JCI Insight. 2024 Feb 22;9(4):e174097. doi: 10.1172/jci.insight.174097. PMID 38271099
- [Derived] Shomaker LB, Tanofsky-Kraff M, Matherne CE, Mehari RD, Olsen CH, Marwitz SE, Bakalar JL, Ranzenhofer LM, Kelly NR, Schvey NA, Burke NL, Cassidy O, Brady SM, Dietz LJ, Wilfley DE, Yanovski SZ, Yanovski JA. A randomized, comparative pilot trial of family-based interpersonal psychotherapy for reducing psychosocial symptoms, disordered-eating, and excess weight gain in at-risk preadolescents with loss-of-control-eating. Int J Eat Disord. 2017 Sep;50(9):1084-1094. doi: 10.1002/eat.22741. Epub 2017 Jul 17. PMID 28714097
- [Derived] Radin RM, Tanofsky-Kraff M, Shomaker LB, Kelly NR, Pickworth CK, Shank LM, Altschul AM, Brady SM, Demidowich AP, Yanovski SZ, Hubbard VS, Yanovski JA. Metabolic characteristics of youth with loss of control eating. Eat Behav. 2015 Dec;19:86-9. doi: 10.1016/j.eatbeh.2015.07.002. Epub 2015 Jul 18. PMID 26210388